CLINICAL TRIAL: NCT04173741
Title: A Correlation Study in the Intensive Care Unit Between the Respiratory Variation Ratios of Internal Jugular Vein and Inferior Vena Cava Before and After Passive Leg Raise
Brief Title: Is There Any Correlation Between Respiratory Variation Ratios of Internal Jugular Vein and Inferior Vena Cava?
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Asli Melek, Principal Investigator, Hacettepe University
Other Study IDs: GO 17/427
Record Dates: First submitted 2019-11-16; First posted 2019-11-22 (Actual); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Critically Ill
Keywords: Positive Pressure Ventilation; Fluid Responsiveness; Passive Leg Raise; Inferior Vena Cava; Internal Jugular Vein; Interobserver Variability; Ultrasound
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Leg Rise Position - 3 Minutes: Patients who stayed in passive leg rise position for 3 minutes
  Interventions: Other: USG measurement
- Leg Rise Position - 1 Minute: Patients who stayed in passive leg rise position for 1 minute
  Interventions: Other: USG measurement

INTERVENTIONS:
Other: USG measurement — IVC was visualized in the subxiphoid long axis by using convex probe (5-1 MHz). Diameters of IVC was measured 2 cm caudally to the junction of hepatic vein in M-mode. IJV diameter was measured in the short axis by using linear probe (12-5 MHz) and M-mode. IJV visualized in the junction of cricothyroid membrane level and midclavicular line. Maximum and minimum diameter values were measured in the M mode. Distensibility (maximum diameter - minimum diameter / minimum diameter) and collapsibility (maximum diameter - minimum diameter / maximum diameter) indices were calculated after USG measurements were done.

SUMMARY:
Intravascular volume assesment is important for the management of the patients in the intensive care unit. Respiratory variation ratio of the inferior vena cava (IVC) can be determined by ultrasonography (USG) and is a useful tool for hemodynamic evaluation of the patient.

Aim of this study is to search for correlation between respiratory variation ratios of the internal jugular vein (IJV) and the IVC before and after passive leg raise. Another aim of this study is to search for variability between ultrasonographic measurements of different doctors.

DETAILED DESCRIPTION:
The investigators measure the internal jugular vein (IJV) diameter in the short axis by using the linear probe (12-5 MHz) and M-mode of the ultrasound device in the junction of cricothyroid membrane level and midclavicular line. The inferior vena cava (IVC) is visualized in the subxiphoid long axis by using the convex probe (5-1 MHz). Diameter of the IVC is measured 2 cm caudally to the junction of the hepatic vein in M-mode. All measurements are done separately by 3 different doctors; one senior anesthesiology resident, one anesthesiology and critical care medicine fellow and one professor in anesthesiology and critical care. The first measurements of the IVC and the IJV are done in the supine position and the second ones are done after passive leg raise. Passive leg raise is done for 1 minute in the first group and for 3 minutes in the second group. Then distensibility (maximum diameter - minimum diameter / minimum diameter) and collapsibility (maximum diameter - minimum diameter / maximum diameter) indices are calculated. No fluid therapy or medication are given to the patients according to these measurements.

Oxygen saturation, hearth rate and blood pressure levels are recorded before and after the measurements. The investigators also record age, gender, weight, height, body mass index, causes of admission, comorbidities, ventilator settings, vasoactive and diuretic medications, fluid intake and output volumes, Acute Physiology and Chronic Health Evaluation II (APACHE II) and Sepsis-Related Organ Failure Assessment (SOFA) scores in the day of admission, Acute Physiology Score (APS) and SOFA scores in the day of measurement and length of stay in the intensive care unit.

Patients with infection or surgical sutures in the site of measurement areas, intraabdominal hypertension, severe aortic regurgitation or lower extremity amputation history are excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated
* Over 18 years of age

Exclusion Criteria:

* Infection in the site of measurement areas
* Surgical sutures in the site of measurement areas
* Intraabdominal hypertension
* Severe aortic regurgitation
* Lower extremity amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients in the intensive care unit over 18 years of age
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asli Melek, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Hospital Anesthesiology Intensive Care Unit, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Nakamura K, Tomida M, Ando T, Sen K, Inokuchi R, Kobayashi E, Nakajima S, Sakuma I, Yahagi N. Cardiac variation of inferior vena cava: new concept in the evaluation of intravascular blood volume. J Med Ultrason (2001). 2013 Jul;40(3):205-9. doi: 10.1007/s10396-013-0435-6. Epub 2013 Feb 27. PMID 27277237
- [Background] Nakamura K, Qian K, Ando T, Inokuchi R, Doi K, Kobayashi E, Sakuma I, Nakajima S, Yahagi N. Cardiac Variation of Internal Jugular Vein for the Evaluation of Hemodynamics. Ultrasound Med Biol. 2016 Aug;42(8):1764-70. doi: 10.1016/j.ultrasmedbio.2016.03.003. Epub 2016 Apr 20. PMID 27108039
- [Background] Akilli NB, Cander B, Dundar ZD, Koylu R. A new parameter for the diagnosis of hemorrhagic shock: jugular index. J Crit Care. 2012 Oct;27(5):530.e13-8. doi: 10.1016/j.jcrc.2012.01.011. Epub 2012 Mar 3. PMID 22386226
- [Background] Preau S, Saulnier F, Dewavrin F, Durocher A, Chagnon JL. Passive leg raising is predictive of fluid responsiveness in spontaneously breathing patients with severe sepsis or acute pancreatitis. Crit Care Med. 2010 Mar;38(3):819-25. doi: 10.1097/CCM.0b013e3181c8fe7a. PMID 20016380

RESULTS

PARTICIPANT FLOW:
Groups:
- Leg Rise Position - 3 Minutes: Patients who stayed in passive leg rise position for 3 minutes
  Ultrasonography (USG) measurement: Inferior vena cava (IVC) was visualized in the subxiphoid long axis by using convex probe (5-1 MHz). Diameters of IVC was measured 2 cm caudally to the junction of hepatic vein in M-mode. Internal jugular vein (IJV) diameter was measured in the short axis by using linear probe (12-5 MHz) and M-mode. IJV visualized in the junction of cricothyroid membrane level and midclavicular line. Maximum and minimum diameter values were measured in the M mode. Distensibility (maximum diameter - minimum diameter / minimum diameter) and collapsibility (maximum diameter - minimum diameter / maximum diameter) indices were calculated after USG measurements were done.
- Leg Rise Position - 1 Minute: Patients who stayed in passive leg rise position for 1 minute
  Ultrasonography (USG) measurement: Inferior vena cava (IVC) was visualized in the subxiphoid long axis by using convex probe (5-1 MHz). Diameters of IVC was measured 2 cm caudally to the junction of hepatic vein in M-mode. Internal jugular vein (IJV) diameter was measured in the short axis by using linear probe (12-5 MHz) and M-mode. IJV visualized in the junction of cricothyroid membrane level and midclavicular line. Maximum and minimum diameter values were measured in the M mode. Distensibility (maximum diameter - minimum diameter / minimum diameter) and collapsibility (maximum diameter - minimum diameter / maximum diameter) indices were calculated after USG measurements were done.
Period: Overall Study
Arm/Group | Leg Rise Position - 3 Minutes | Leg Rise Position - 1 Minute
Started | 23 | 23
Completed | 22 | 22
Not Completed | 1 | 1
Not completed — IVC measurement cannot be done | 1 | 1

BASELINE CHARACTERISTICS:
Population: IVC cannot be visualized by any of the physicians in 1 patient in Group A and in 1 patient in Group B. Statistical analysis is done with total of 44 patients.
Groups:
- Group A: Patients who stayed in passive leg rise position for 3 minutes
  USG measurement: IVC was visualized in the subxiphoid long axis by using convex probe (5-1 MHz). Diameters of IVC was measured 2 cm caudally to the junction of hepatic vein in M-mode. IJV diameter was measured in the short axis by using linear probe (12-5 MHz) and M-mode. IJV visualized in the junction of cricothyroid membrane level and midclavicular line. Maximum and minimum diameter values were measured in the M mode. Distensibility (maximum diameter - minimum diameter / minimum diameter) and collapsibility (maximum diameter - minimum diameter / maximum diameter) indices were calculated after USG measurements were done.
- Group B: Patients who stayed in passive leg rise position for 1 minute
  USG measurement: IVC was visualized in the subxiphoid long axis by using convex probe (5-1 MHz). Diameters of IVC was measured 2 cm caudally to the junction of hepatic vein in M-mode. IJV diameter was measured in the short axis by using linear probe (12-5 MHz) and M-mode. IJV visualized in the junction of cricothyroid membrane level and midclavicular line. Maximum and minimum diameter values were measured in the M mode. Distensibility (maximum diameter - minimum diameter / minimum diameter) and collapsibility (maximum diameter - minimum diameter / maximum diameter) indices were calculated after USG measurements were done.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Median (Full Range); unit: years] | 66 [19 to 95] | 74 [21 to 94] | 71 [19 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 10 | 11 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Ultrasonography (USG) Measurements
Description: Because of the medium-high interrater correlation between USG measurements of the physicians, statistical analysis were done with the mean of USG measurements of 3 doctors.
Time Frame: through study completion, 3 days
Measure: Median (Full Range); unit: centimeter
Groups:
- Leg Rise Position - 3 Minutes: Patients who stayed in passive leg rise position for 3 minutes
  Ultrasonography (USG) measurement: Inferior vena cava (IVC) was visualized in the subxiphoid long axis by using convex probe (5-1 MHz). Diameters of IVC was measured 2 cm caudally to the junction of hepatic vein in M-mode. IJV diameter was measured in the short axis by using linear probe (12-5 MHz) and M-mode. Internal jugular vein (IJV) visualized in the junction of cricothyroid membrane level and midclavicular line. Maximum and minimum diameter values were measured in the M mode. Distensibility (maximum diameter - minimum diameter / minimum diameter) and collapsibility (maximum diameter - minimum diameter / maximum diameter) indices were calculated after USG measurements were done.
- Leg Rise Position - 1 Minute: Patients who stayed in passive leg rise position for 1 minute
  Ultrasonography (USG) measurement: Inferior vena cava (IVC) was visualized in the subxiphoid long axis by using convex probe (5-1 MHz). Diameters of IVC was measured 2 cm caudally to the junction of hepatic vein in M-mode. IJV diameter was measured in the short axis by using linear probe (12-5 MHz) and M-mode. Internal jugular vein (IJV) visualized in the junction of cricothyroid membrane level and midclavicular line. Maximum and minimum diameter values were measured in the M mode. Distensibility (maximum diameter - minimum diameter / minimum diameter) and collapsibility (maximum diameter - minimum diameter / maximum diameter) indices were calculated after USG measurements were done.
Arm/Group | Leg Rise Position - 3 Minutes | Leg Rise Position - 1 Minute
Number analyzed (Participants) | 22 | 22
centimeter
  Maximum diameter of IVC in supine position | 1.80 [0.98 to 2.53] | 1.97 [1.26 to 2.60]
  Minimum diameter of IVC in supine position | 1.22 [0.14 to 2.14] | 1.61 [0.33 to 2.32]
  Maximum diameter of IVC after passive leg raise | 1.75 [0.84 to 2.83] | 2.13 [1.26 to 2.88]
  Minimum diameter of IVC after passive leg raise | 1.33 [0.26 to 2.52] | 1.67 [0.44 to 2.51]
  Maximum diameter of IJV in supine position | 1.03 [0.51 to 1.54] | 1.06 [0.45 to 1.52]
  Minimum diameter of IJV in supine position | 0.91 [0.27 to 1.41] | 0.89 [0.31 to 1.29]
  Maximum diameter of IJV after passive leg raise | 1.08 [0.47 to 1.52] | 1.00 [0.42 to 1.64]
  Minimum diameter of IJV after passive leg raise | 0.90 [0.41 to 1.47] | 0.85 [0.33 to 1.28]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 month.
Description: Only All-Cause Mortality were assessed. Serious and Other (Not Including Serious) Adverse Events were not assessed.
Arm/Group | Leg Rise Position - 3 Minutes | Leg Rise Position - 1 Minute
All-Cause Mortality (participants affected / at risk) | 9/23 | 12/23
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT04173741/Prot_SAP_000.pdf